CLINICAL TRIAL: NCT03389672
Title: a Modified Method That Improved Residency Neuraxial Anesthesia Performance and Reduced Patient Complications
Brief Title: Modified Paramedian Versus Conventional Technique in the Residency Training: An Observational Study
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB200812040R
Record Dates: First submitted 2017-12-26; First posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2011-01

CONDITIONS: Anesthesia
Keywords: patient safety; residency training
MeSH Terms: interventions — Anesthesia, Spinal; Anesthesia, Epidural

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- spinal anesthesia: The anesthesia technique were applied with modified approach and conventional approach
  Interventions: Procedure: spinal anesthesia
- epidural anesthesia: The anesthesia technique were applied with modified approach and conventional approach
  Interventions: Procedure: epidural anesthesia
- combined spinal-epidural anesthesia: The anesthesia technique were applied with modified approach and conventional approach
  Interventions: Procedure: combined spinal-epidural anesthesia

INTERVENTIONS:
Procedure: spinal anesthesia — For conventional spinal anesthesia, injection site was 1 cm lateral and 1 cm caudal to the spinous process, and the needle was directed cephalad and medially to the epidural-subarachnoid space by the operator. For modified method, we reduced the distance from 1cm to 0.5cm in each directions.
  Groups: spinal anesthesia
Procedure: epidural anesthesia — For conventional epidural anesthesia, injection site was 1 cm lateral and 1 cm caudal to the spinous process, and the needle was directed cephalad and medially to the epidural-subarachnoid space by the operator. For modified method, we reduced the distance from 1cm to 0.5cm in each directions.
  Groups: epidural anesthesia
Procedure: combined spinal-epidural anesthesia — For conventional combined spinal-epidural anesthesia, injection site was 1 cm lateral and 1 cm caudal to the spinous process, and the needle was directed cephalad and medially to the epidural-subarachnoid space by the operator. For modified method, we reduced the distance from 1cm to 0.5cm in each directions.
  Groups: combined spinal-epidural anesthesia

SUMMARY:
Residency training includes positive and negative aspects. Well-trained doctors must be educated, but the process may bring additional risks to patients. Anesthesiologists' performance when conducting neuraxial anesthesia is related to their experience. We hypothesized that a modified neuraxial anesthesia method would improve both residency training and patient safety.

DETAILED DESCRIPTION:
Residency training is performed using trial and error. Several studies have shown that the training process, practice period, and resident's attitude are important factors for determining performance. During the training process, neuraxial anesthesia safety is related to the operator's experience. Ultrasound can improve resident performance; however, using ultrasound technologies in well-established training programs may not be practical for all residencies.

The paramedian approach bypasses most of the bony structures that may impede the advancement of an epidural needle in the midline approach. However, the paramedian approach requires a sharpened three-dimensional insight compared with the midline approach. We hypothesized that the higher the three-dimensional barrier, the higher the complications and number of puncture attempts. A modified paramedian approach may improve residency training and patient safety. The aim of this study was to investigate whether the modified method decreased practice attempts and patient complications.

ELIGIBILITY:
Inclusion Criteria:

* parturients who were elective for cesarean section

Exclusion Criteria:

* history of allergy to the medications used in this study
* chronic or acute headaches
* possible conversion to general anesthesia
* other contraindications to practice (infection, coagulopathy, abnormal spinal anatomy, unstable vital signs, and refusal to participate in the study)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — parturients who were elective for cesarean section
Study Population: All parturients received regional anesthesia in the decubitus position, and the procedures were performed in the L3-4 or L4-5 interspace. For the conventional method, the injection site was 1 cm lateral and 1 cm caudal to the spinous process, and the needle was directed cephalad and medially to the epidural-subarachnoid space by the operator. For the modified method, the injection site was 0.5 cm lateral and 0.5 cm caudal to the spinous process, and the process was the same as the conventional method
Sampling Method: Non-Probability Sample
Enrollment: 518 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2012-09-30 (Actual); Study Completion 2012-09-30 (Actual)

PRIMARY OUTCOMES:
attempts | at least three days
  the number of skin-to-site needle punctures

SECONDARY OUTCOMES:
complication | at least three days
  all types of complications, including a post dura-puncture headache epidural hematoma, infection, or any unexpected neurologic injury

CONTACTS AND LOCATIONS:
Overall Officials: Hong-Nerng Ho, PhD, Study Chair — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request

REFERENCES:
- [Background] Ambardekar AP. Selecting anesthesiology residency candidates-Beyond the numbers. J Clin Anesth. 2017 Sep;41:38-39. doi: 10.1016/j.jclinane.2017.05.006. No abstract available. PMID 28802600
- [Background] de Oliveira Filho GR. The construction of learning curves for basic skills in anesthetic procedures: an application for the cumulative sum method. Anesth Analg. 2002 Aug;95(2):411-6, table of contents. doi: 10.1097/00000539-200208000-00033. PMID 12145063
- [Background] Martin G, Lineberger CK, MacLeod DB, El-Moalem HE, Breslin DS, Hardman D, D'Ercole F. A new teaching model for resident training in regional anesthesia. Anesth Analg. 2002 Nov;95(5):1423-7, table of contents. doi: 10.1097/00000539-200211000-00059. PMID 12401637
- [Background] Sahin T, Balaban O, Sahin L, Solak M, Toker K. A randomized controlled trial of preinsertion ultrasound guidance for spinal anaesthesia in pregnancy: outcomes among obese and lean parturients: ultrasound for spinal anesthesia in pregnancy. J Anesth. 2014 Jun;28(3):413-9. doi: 10.1007/s00540-013-1726-1. Epub 2013 Oct 20. PMID 24141882
- [Background] Shaikh F, Brzezinski J, Alexander S, Arzola C, Carvalho JC, Beyene J, Sung L. Ultrasound imaging for lumbar punctures and epidural catheterisations: systematic review and meta-analysis. BMJ. 2013 Mar 26;346:f1720. doi: 10.1136/bmj.f1720. PMID 23532866
- [Background] Perlas A, Chaparro LE, Chin KJ. Lumbar Neuraxial Ultrasound for Spinal and Epidural Anesthesia: A Systematic Review and Meta-Analysis. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):251-60. doi: 10.1097/AAP.0000000000000184. PMID 25493689
- [Background] Vallejo MC, Phelps AL, Singh S, Orebaugh SL, Sah N. Ultrasound decreases the failed labor epidural rate in resident trainees. Int J Obstet Anesth. 2010 Oct;19(4):373-8. doi: 10.1016/j.ijoa.2010.04.002. Epub 2010 Aug 8. PMID 20696564
- [Derived] Chen SH, Chen SS, Lai CL, Su FY, Tzeng IS, Chen LK. Modified paramedian versus conventional paramedian technique in the residency training: an observational study. BMC Med Educ. 2020 Jul 2;20(1):211. doi: 10.1186/s12909-020-02118-0. PMID 32615968